CLINICAL TRIAL: NCT03674411
Title: Single-Arm, Open Label, Interventional Phase II Clinical Trial Evaluating MGTA-456 in Patients With High-Risk Malignancy
Brief Title: Trial Evaluating MGTA-456 in Patients With High-Risk Malignancy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018LS051; MT2018-06 (Other: University of Minnesota Masonic Cancer Center)
Record Dates: First submitted 2018-09-14; First posted 2018-09-17 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphocytic Leukemia; Biphenotypic/Undifferentiated Leukemia; Chronic Myelogenous Leukemia; Myelodysplasia; Relapsed Large Cell Lymphoma; Mantle Cell Lymphoma; Hodgkin Lymphoma; Burkitt Lymphoma; Relapsed T-Cell Lymphoma; Lymphoplasmacytic Lymphoma
Keywords: AML; ALL; CML; MCL
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Anemia, Refractory, with Excess of Blasts; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Hodgkin Disease; Burkitt Lymphoma; Lymphoma, T-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — fludarabine; Cyclophosphamide; Whole-Body Irradiation; Tacrolimus; Triamcinolone; Mycophenolic Acid; Granulocyte Colony-Stimulating Factor; Busulfan; Melphalan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- FLU, CY, TBI + MGTA-456 infusion (Experimental): All patients will receive MGTA-456 on the day of transplantation after myeloablative conditioning.
  All patients aged 3-55 years will be conditioned with cyclophosphamide (CY) 120 mg/kg total dose, fludarabine (FLU) 75 m/m2 total dose and total body irradiation (TBI) 1320 cGy total dose as well as tacrolimus (Tac) and mycophenolate mofetil (MMF) immunoprophylaxis and granulocyte-colony stimulating factor (G-CSF)
  Interventions: Drug: Fludarabine (FLU); Drug: Cyclophosphamide (CY); Drug: Total Body Irradiation (TBI); Drug: Tacrolimus (Tac); Drug: Mycophenolate Mofetil (MMF); Drug: Granulocyte Colony-Stimulating Factor (G-CSF); Drug: MGTA 456 Infusion
- BU,FLU, MEL + MGTA-456 infusion (Experimental): All young children <3 years of age at the time of diagnosis will receive MGTA-456 on the day of transplantation after a non-TBI containing myeloablative conditioning as TBI may have a damaging effect on brain development in the very young child. All patients aged 0-3 years will be conditioned with busulfan (BU), FLU and melphalan (MEL) as well as Tac/MMF immunoprophylaxis and G-CSF
  Interventions: Drug: Fludarabine (FLU); Drug: Mycophenolate Mofetil (MMF); Drug: Granulocyte Colony-Stimulating Factor (G-CSF); Drug: Busulfan (BU); Drug: Melphalan; Drug: MGTA 456 Infusion

INTERVENTIONS:
Drug: Fludarabine (FLU) — 25 mg/m2 IV over 1 hour (<10 kg: 0.83 mg/kg IV over 1 hour)
Drug: Cyclophosphamide (CY) — 60 mg/kg IV over 2 hours
  Arms: FLU, CY, TBI + MGTA-456 infusion
Drug: Total Body Irradiation (TBI) — 165 cGy twice daily
  Arms: FLU, CY, TBI + MGTA-456 infusion
Drug: Tacrolimus (Tac) — Tacrolimus will start day -3 and will be administered as a continuous IV infusion at a starting dose of 0.03 mg/kg/day. Goal trough levels will be 10-15 ng/mL for the first 14 days post-transplant and then decreased to a goal of 5-10 ng/ml thereafter.
  Arms: FLU, CY, TBI + MGTA-456 infusion
Drug: Mycophenolate Mofetil (MMF) — MMF 3 gram/day IV/PO for adult patients divided in 2 or 3 doses. Pediatric patients will receive MMF at the dose of 15 mg/kg/dose (max 1 gram per dose) every 8 hours beginning day -3.
Drug: Granulocyte Colony-Stimulating Factor (G-CSF) — 5 ug/kg/d until the absolute neutrophil count (ANC) is >2500/uL for 2 consecutive days
Drug: Busulfan (BU) — BU IV once daily with dose based on Pharmacokinetics (PK) calculator over 3 hours
  Arms: BU,FLU, MEL + MGTA-456 infusion
Drug: Melphalan — 50 mg/m2/day (1.7 mg/kg/day if < 10 kg) IV over 30 min
  Arms: BU,FLU, MEL + MGTA-456 infusion
Drug: MGTA 456 Infusion — The target cell dose is >10 x 106 CD34/kg with a maximum TNC 2.7 x 108/kg for children (<18 years) and 8.1 × 108 cells/kg [expanded product only] for adults based on the highest cell dose windows evaluated in prior studies.

SUMMARY:
This is an single arm, open label, interventional phase II trial evaluating the efficacy of umbilical cord blood (UCB) hematopoietic stem and progenitor cells (HSPC) expanded in culture with stimulatory cytokines (SCF, Flt-3L, IL-6 and thromopoietin) on lympho-hematopoietic recovery. Patients will receive a uniform myeloablative conditioning and post-transplant immunoprophylaxis.

ELIGIBILITY:
Age, Unit Cell Dose and HLA Match Criteria

* Subjects must be ≤55 years of age
* Subjects must weigh >11 kg
* Subjects must have a partially HLA matched UCB unit with a pre-cryopreserved TNC dose >1.0 x 107 per kilogram recipient weight. HLA matching is initially based on a minimum of 5 of 8 HLA alleles at high resolution A, B, C, DRB1 typing; searches will be performed according to the current Magenta Cord Blood Search Algorithm.

Eligible Diseases:

* Acute myelogenous leukemia (AML) in morphological complete remission with:

  * Minimal residual disease (MRD) by flow cytometry, or
  * Intermediate to high risk leukemia in first (CR1) based on institutional criteria, eg. not favorable risk AML which is defined as having one of the following:

    * t(8,21) without cKIT mutation
    * inv(16) or t(16;16) without cKIT mutation
    * Normal karyotype with mutated NPM1 but FLT3-ITD wild type
    * Normal karyotype with double mutated CEBPA
    * Acute promyelocytic leukemia (APL) in first molecular remission at the end of consolidation
  * Any second or subsequent CR, or
  * Secondary AML with prior malignancy that has been in remission for at least 12 months.

    * Acute lymphocytic leukemia (ALL) at the following stages:
    * High risk first morphological, cytogenetic and molecular CR with:

      * MRD by flow cytometry, or
      * Diagnosis of Philadelphia chromosome (Ph)+ ALL, or
      * MLL rearrangement at diagnosis with slow early response at Day 14, or
      * Hypodiploidy (< 44 chromosomes or DNA index < 0.81) at diagnosis, or
      * End of induction M3 bone marrow, or
      * End of induction M2 with M2-3 at Day 42.
    * High risk second CR based on institutional criteria (eg, for children, bone marrow relapse <36 months from induction or T-lineage bone marrow relapse or very early isolated central nervous system (CNS) relapse <6 months from diagnosis, or slow re-induction (stage M2-3 at day 28 after induction) regardless of length remission. All patients with MRD by flow cytometry.
    * Any third or subsequent CR.
  * Secondary ALL
  * Biphenotypic/undifferentiated leukemia in morphological, cytogenetic and molecular CR .
  * Chronic Myelogenous Leukemia (CML) in high risk first chronic phase (failure of two tyrosine kinase inhibitors (TKI) or TKI intolerance), accelerated phase or second chronic phase.
  * Myelodysplasia (MDS) IPSS Int-2 or High risk (i.e. RAEB, RAEBt <5% blasts) or other high risk features, including multiple cytopenias, high risk cytogenetics or lack of response to standard therapy..
  * Relapsed large-cell lymphoma, mantle-cell lymphoma and Hodgkin lymphoma that is chemotherapy sensitive and ineligible for an autologous transplant.
  * Burkitt's lymphoma in CR2 or subsequent CR.
  * Relapsed T-cell lymphoma that is chemotherapy sensitive in CR/PR that is ineligible for an autologous transplant.

Organ Specific Inclusion Criteria

* Karnofsky score ≥70 (16 years and older), Lansky play score >50 (children 2-16 years, or 'adequate' score for children <2 years, as detailed in Appendix II.
* Adequate organ function defined as:

  * Renal: Serum creatinine within normal range for age, or if serum creatinine outside normal range for age, then creatinine clearance >40 ml/min or GFR ≥70 mL/min/1.73 m2.normal for age
  * Hepatic: Bilirubin <3x upper limit of normal (ULN) and AST, ALT and alkaline phosphatase <5x ULN.
  * Pulmonary function: DLCO, FEV1, FEC (diffusion capacity) >5030% of predicted (corrected for hemoglobin); if unable to perform pulmonary function tests, then O2 saturation >95% on room air.
* Cardiac: No uncontrolled arrhythmia and left ventricular ejection fraction at rest must be >3545%.
* Available 'back-up' HSPC graft (e.g, second UCB unit, haploidentical related donor).
* Females of child bearing potential and sexually active males must agree to use adequate birth control during study treatment.
* Voluntary written consent signed (adult or parental) before performance of any study-related procedure not part of normal medical care.

Exclusion Criteria

* Patients with a HLA matched sibling donor or a HLA matched unrelated donor who is available for marrow or peripheral blood stem cell collection at the desired time of transplant.
* Pregnant or breast feeding. The agents used in this study may be teratogenic to a fetus and there is no information on the excretion of agents into breast milk. Females of childbearing potential must have a blood test or urine study within 14 days prior to study enrollment to rule out pregnancy.
* Evidence of human immunodeficiency virus (HIV) infection or known HIV positive serology.
* Active bacterial, viral or fungal infection (currently taking medication and persistence of clinical signs and symptoms) with a minimum of 4 weeks of anti-fungal treatment
* Prior autologous or allogeneic transplant.
* Other active malignancy.
* Subjects >2 3 years of age unable to receive TBI 1320 cGy due to extensive prior therapy including >12 months alkylator therapy or >6 months alkylator therapy with extensive radiation, or prior Y-90 ibritumomab (Zevalin) or I-131 tostumomab (Bexxar), as part of their salvage therapy.

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2026-12-01 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- FLU, CY, TBI + MGTA-456 Infusion: All patients aged 3-55 years will be conditioned with cyclophosphamide (CY) 120 mg/kg total dose, fludarabine (FLU) 75 m/m2 total dose and total body irradiation (TBI) 1320 cGy total dose as well as tacrolimus (Tac) and mycophenolate mofetil (MMF) immunoprophylaxis and granulocyte-colony stimulating factor (G-CSF)
Period: Overall Study
Arm/Group | FLU, CY, TBI + MGTA-456 Infusion | BU,FLU, MEL + MGTA-456 Infusion
Started | 20 | 2
Completed | 16 | 2
Not Completed | 4 | 0
Not completed — Non-treatment | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FLU, CY, TBI + MGTA-456 Infusion | BU,FLU, MEL + MGTA-456 Infusion | Total
Number analyzed (Participants) | 16 | 2 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 2 | 7
  Between 18 and 65 years | 11 | 0 | 11
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 11 | 1 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 13 | 2 | 15
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 10 | 0 | 10
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 16 | 2 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Neutrophil Recover
Description: Percentage of participants with neutrophil recovery by day 14 after transplantation in recipients of MGTA-456.
Time Frame: Day 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FLU, CY, TBI + MGTA-456 Infusion | BU,FLU, MEL + MGTA-456 Infusion
Number analyzed (Participants) | 16 | 2
Percentage of participants | 31 [14 to 60] | 50 [9 to 99]

2. Secondary Outcome: Number of Days Alive Without Hospitalization
Description: Number of days alive without hospitalization between days 0 and 100 after transplantation
Time Frame: Day 0 and Day 100
Measure: Median (Full Range); unit: Days
Arm/Group | FLU, CY, TBI + MGTA-456 Infusion | BU,FLU, MEL + MGTA-456 Infusion
Number analyzed (Participants) | 16 | 2
Days | 67.5 [18 to 85] | 33 [0 to 66]

3. Secondary Outcome: Secondary Graft Failure
Description: Incidence of secondary graft failure
Time Frame: 2 Years
Measure: Number; unit: Percentage of participants
Arm/Group | FLU, CY, TBI + MGTA-456 Infusion | BU,FLU, MEL + MGTA-456 Infusion
Number analyzed (Participants) | 16 | 2
Percentage of participants | 37.5 | 0

4. Secondary Outcome: Platelet Recovery
Description: Incidence of platelet recovery at day 42
Time Frame: Day 42
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FLU, CY, TBI + MGTA-456 Infusion | BU,FLU, MEL + MGTA-456 Infusion
Number analyzed (Participants) | 16 | 2
Percentage of participants | 56 [33 to 80] | 50 [1 to 99]

5. Secondary Outcome: Treatment Related Mortality (TRM)
Description: Incidence of TRM at 6 months
Time Frame: 6 Months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FLU, CY, TBI + MGTA-456 Infusion | BU,FLU, MEL + MGTA-456 Infusion
Number analyzed (Participants) | 16 | 2
Percentage of participants | 6 [0 to 18] | 50 [15 to 85]

6. Secondary Outcome: Grades II-IV Acute GVHD
Description: Incidence of grades II-IV acute GVHD at day 100
Time Frame: Day 100
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FLU, CY, TBI + MGTA-456 Infusion | BU,FLU, MEL + MGTA-456 Infusion
Number analyzed (Participants) | 16 | 2
Percentage of participants | 25 [4 to 46] | 0 [0 to 100]

7. Secondary Outcome: Grades III-IV Acute GVHD
Description: Incidence of grades III-IV acute GVHD at day 100
Time Frame: Day 100
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FLU, CY, TBI + MGTA-456 Infusion | BU,FLU, MEL + MGTA-456 Infusion
Number analyzed (Participants) | 16 | 2
Percentage of participants | 19 [0 to 37] | 0 [0 to 100]

8. Secondary Outcome: Chronic GVHD
Description: Incidence of chronic GVHD at 1 year
Time Frame: 1 Year
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FLU, CY, TBI + MGTA-456 Infusion | BU,FLU, MEL + MGTA-456 Infusion
Number analyzed (Participants) | 16 | 2
Percentage of participants | 13 [0 to 28] | 0 [0 to 100]

9. Secondary Outcome: Relapse
Description: Incidence of relapse at 2 years
Time Frame: 2 Years
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FLU, CY, TBI + MGTA-456 Infusion | BU,FLU, MEL + MGTA-456 Infusion
Number analyzed (Participants) | 16 | 2
Percentage of participants | 25 [4 to 46] | 50 [1 to 99]

10. Secondary Outcome: Non-catheter Associated Bacterial Infections
Description: Incidence of non-catheter associated bacterial infections by day 100
Time Frame: Day 100
Measure: Number; unit: Percentage of participants
Arm/Group | FLU, CY, TBI + MGTA-456 Infusion | BU,FLU, MEL + MGTA-456 Infusion
Number analyzed (Participants) | 16 | 2
Percentage of participants | 6 | 0

11. Secondary Outcome: Overall Survival (OS)
Description: Incidence of overall survival (OS) at 2 years
Time Frame: 2 Years
Measure: Number; unit: Percentage of participants
Arm/Group | FLU, CY, TBI + MGTA-456 Infusion | BU,FLU, MEL + MGTA-456 Infusion
Number analyzed (Participants) | 16 | 2
Percentage of participants | 69 | 0

12. Secondary Outcome: Event-Free Survival (EFS)
Description: Incidence of event-free survival (EFS) at 2 years
Time Frame: 2 Years
Measure: Number; unit: Percentage of participants
Arm/Group | FLU, CY, TBI + MGTA-456 Infusion | BU,FLU, MEL + MGTA-456 Infusion
Number analyzed (Participants) | 16 | 2
Percentage of participants | 69 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | FLU, CY, TBI + MGTA-456 Infusion | BU,FLU, MEL + MGTA-456 Infusion
All-Cause Mortality (participants affected / at risk) | 5/16 | 2/2
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/2
Other Adverse Events (participants affected / at risk) | 0/16 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/11/NCT03674411/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/11/NCT03674411/ICF_001.pdf